CLINICAL TRIAL: NCT05261776
Title: The Effects of Pilates on Functional Capacity and Blood Glucose Levels in Adults With Diabetes Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00240
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: glycemic control; hyperglycemia; functionality; Pilates exercises
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as accessor of the study would be kept blind of the treatment group to which patient would be allocated. After the complete initial screening process, every recruited patient will be accessed by an independent assessor, expert will use outcome measuring tools. his will be recorded as baseline measurement assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Experimental): Group-A will receive pilates exercise and standard care
  Interventions: Other: pilates exercise
- Group-B (Active Comparator): Group-B will receive brisk walk and standard care
  Interventions: Other: brisk walk

INTERVENTIONS:
Other: pilates exercise — Pilates exercise for 40 minutes (5 minutes for warm-up and 30 minutes of pilates and 5 minutes for cool down). These participants will continue their standard care.
  Patients in Group-A will get 40 minutes of session, Alternative three days/ week for 12 weeks.
  Arms: Group-A
Other: brisk walk — Brisk walk on treadmill for 40 minutes (5 minutes for warm-up and 30 minutes of brisk walk on treadmill and 5 minutes for cool down). These participants will continue their standard care.
  Patients in Group-B of 40 minutes of session, Alternative three days/ week for 12 weeks.
  Arms: Group-B

SUMMARY:
The aim of this study is to investigate the effects of the Pilates training on Functional Capacity among adults with type 2 diabetes The aim of this study is to investigate the effects of the Pilates training on blood glucose response among adults with type 2 diabetes

DETAILED DESCRIPTION:
A Randomized Control Trial study of 3 month period will be arranged, at Riphah International University Faisalabad after the approval of synopsis. The convenience sampling technique will be selected for registration of patients. According to specified inclusion, exclusion criteria, patients will be chosen. Calculation of Sample size for the study tells need of both males and females (45 yrs-65 yrs) that will fulfill the certain criteria. The participants of group A will receive Pilates exercise and standard care and participants of group B will receive a brisk walk on treadmill and standard care. The evaluation of patients will be done at baseline, at 6th week, 12th week and at follow up after one month of discontinuation of treatment. The patient's outcome will be measured by 6-Minute Walk Test (distance), hemoglobin A1c level and Blood Glucose level and the recording of the patient's data will be at pre-treatment and post-treatment. The data of before treatment and after treatment will be compared at follow up after one month of discontinuation of treatment. For each patient informed consent will be taken. Through Statistical Package of Social Sciences 20 software, data entry and analysis will be done

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patient both male and female with diagnosed with type ii diabetes
* 45-65 years old
* Lack of psychic disease, dementia and mental retardation

Exclusion Criteria:

* ulcers in extremities
* Peripheral neuropathy
* Severe or decompensated heart disease
* Limited coronary heart disease
* Insulin therapy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 12th week
  functional capacity is checked by 6-minute walk test
HbA1c | 12th week
  A hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin.
Blood glucose level | 12th week
  The blood glucose level is the amount of glucose in the blood. Glucose is a sugar that comes from the foods we eat, and it's also formed and stored inside the body

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Zolfaghari N, Faramarzi M, Afkhami-Ardekani M, Afkhami-Ardekani A, Jam Ashkezari S. The Effect of Eight Weeks Pilates Exercise on Testosterone and Sex Hormone Biding Globulin (SHBG) in Women with Type 2 Diabetes. Iranian Journal of Diabetes and Obesity. 2015;7(2):45-9.
- [Background] Dendup T, Feng X, Clingan S, Astell-Burt T. Environmental Risk Factors for Developing Type 2 Diabetes Mellitus: A Systematic Review. Int J Environ Res Public Health. 2018 Jan 5;15(1):78. doi: 10.3390/ijerph15010078. PMID 29304014
- [Background] Silva EFF, Ferreira CMM, Pinho L. Risk factors and complications in type 2 diabetes outpatients. Rev Assoc Med Bras (1992). 2017 Jul;63(7):621-627. doi: 10.1590/1806-9282.63.07.621. PMID 28977088
- [Background] Melo KCB, Araujo FS, Cordeiro Junior CCM, de Andrade KTP, Moreira SR. Pilates Method Training: Functional and Blood Glucose Responses of Older Women With Type 2 Diabetes. J Strength Cond Res. 2020 Apr;34(4):1001-1007. doi: 10.1519/JSC.0000000000002704. PMID 29985228
- [Background] Nomura T, Kawae T, Kataoka H, Ikeda Y. Aging, physical activity, and diabetic complications related to loss of muscle strength in patients with type 2 diabetes. Phys Ther Res. 2018 Nov 30;21(2):33-38. doi: 10.1298/ptr.R0002. eCollection 2018. PMID 30697507
- [Background] Colak TK, Acar G, Dereli EE, Ozgul B, Demirbuken I, Alkac C, Polat MG. Association between the physical activity level and the quality of life of patients with type 2 diabetes mellitus. J Phys Ther Sci. 2016 Jan;28(1):142-7. doi: 10.1589/jpts.28.142. Epub 2016 Jan 30. PMID 26957746
- [Background] 7. Torabian M, Taghadosi M, Ajorpaz NM, Khorasanifar L. The effect of Pilates exercises on general health in women with type 2 diabetes. Life Sci J. 2013;2:1-39.
- [Background] 9. NESREEN G, YASMIN M, HAKEM M, SALLY A. Effect of Pilates Exercise on Cardio Metabolic Risk Factors in Women with Type 2 Diabetes. The Medical Journal of Cairo University. 2019;87(March):851-.
- [Background] 10. Yucel H, Uysal O. Pilates-based mat exercises and parameters of quality of life in women with Type 2 diabetes. Iranian Red Crescent Medical Journal. 2018;20(S1).
- [Background] 11. Hassani N, Heravi-Karimooi M, Rejeh N, Ashtiani MHD, Sharifnia H, Ghanbari M, et al. The effect of pilates exercise on quality of life of elderly women with type 2 diabetes. Payesh (Health Monitor). 2018;17(5):531-9.
- [Background] 12. Mir E, Fathi M. Changes in Plasma Visfatin and Insulin Resistance Index in Obese Women with Type 2 Diabetes after Pilates Exercise. Journal of Health and Care. 2018;20(1):30-9.
- [Background] 13. Sharma D, Kaur J, Rani M, Bansal A, Malik M, Kulandaivelan S. Efficacy of Pilates based mat exercise on quality of life, quality of sleep and satisfaction with life in type 2 diabetes mellitus. Romanian Journal of Diabetes Nutrition and Metabolic Diseases. 2018;25(2):149-56.
- [Background] 14. Zolfaghari N, Faramarzi M, Afkhami-Ardekani M, Afkhami-Ardekani A, Jam Ashkezari S. The Effect of Eight Weeks Pilates Exercise on Testosterone and Sex Hormone Biding Globulin (SHBG) in Women with Type 2 Diabetes. Iranian Journal of Diabetes and Obesity. 2015;7(2):45-9.
- [Background] 15. Ebrahimi F, Mahdavinejad R, Jalily H. The effects of selected Pilates exercises on muscle strength, balance and HbA1c in female patients with diabetes type 2. Journal of Exercise Science and Medicine. 2015;7(2):251-65.